CLINICAL TRIAL: NCT01947270
Title: OPMED STUDY: Multidisciplinary Program "Optimization of Drug Prescription" : Impact on the Quality of Drug Prescription in Hospitalized Elderly Patients
Brief Title: Multidisciplinary Program "Optimization of Drug Prescription" : Impact on the Quality of Drug Prescription in Hospitalized Elderly Patients
Acronym: OPMED
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50789
Record Dates: First submitted 2013-07-26; First posted 2013-09-20 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Potentially Inappropriate Medications
Keywords: Potentially inappropriate medications; Elderly; Prevention; Multidisciplinary program; Checklist; Stepped wedge design; AGED, 75 AND OVER

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Patients of this group are hospitalized in a time frame where the multidisciplinary intervention program is not implemented in the medical department. Drug prescriptions are conducted under usual care in the department.
- Intervention group: Patients of this group are hospitalized in a time frame where the multidisciplinary intervention program is implemented in the medical department.
  Interventions: Other: " Optimisation de la Prescription MEDicamenteuse " ("Optimization of drug prescribing")

INTERVENTIONS:
Other: " Optimisation de la Prescription MEDicamenteuse " ("Optimization of drug prescribing") — The multidisciplinary intervention program include:
  * Awareness and training of doctors by two experts (a geriatrician and a pharmacist) within participating departments.
  * Implementation of a checklist which aims to conduct an adapted and standardized pharmaceutical analysis
  Groups: Intervention group

SUMMARY:
Drug prescription is a fundamental component of care for the elderly. Even if drugs are a chance for the older patient, because of changes in pharmacological, pharmacokinetic and pharmacodynamic parameters related with age and acute/or chronic pathologies, the risks associated with drug prescription, particularly those associated with potentially inappropriate medication (PIM), are increased in the elderly.

We suppose that many of hospitalized elderly have at least one prescribed medication without valid indication. Conversely, many diseases are currently undertreated in elderly patients: e.g. medicines used to treat heart failure and osteoporosis are underused in 20 to 70% of patients. Moreover, PMI prescription is associated with an increased of morbidity, mortality, risk of drug-related adverse events, utilization of health care system, care costs and impairment of quality of life. Thus, optimization of drug prescription is a major concern for improvement of the quality and safety of care in elderly.

The investigators' hypothesis is that a multidisciplinary program entitled "Optimisation de la Prescription MEDicamenteuse" ("Optimization of drug prescribing") focused on drug prescription optimization including a physician training to the specificity of the drug prescription in the elderly and a checklist allowing an adapted and standardized pharmaceutical analysis is effective in reducing PIM in elderly patients hospitalized in short-term medical and geriatric care departments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged over 75 years hospitalized in one of the participating department
* Patient agreed to participate

Exclusion Criteria:

* Patient with a predictive length of stay equal or less than 48 hours
* Patients admitted in terminal illness

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized elderly patients from 75 years old.
Sampling Method: Non-Probability Sample
Enrollment: 3055 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of potentially inappropriate medications (PIM) prescribed in discharge of hospitalized patients from 75 years old. | at discharge (average 3 weeks)
  Proportion of prescribed PIM will be expressed as the ratio of PIM to the total number of medication in discharge prescription sheet.
  PIM will be identified by 2 experts (1 doctor and 1 pharmacist) based on criteria from the lists STOPP/START and Laroche.

SECONDARY OUTCOMES:
Total number of drugs prescribed per discharge prescription sheet | at discharge (average 3 weeks)
Number of rehospitalization within 12 months following discharge | 12 months after inclusion
Number of emergency admission within 12 months following hospitalization | 12 months after inclusion
Mortality within 12 months after hospitalization | 12 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon, France